CLINICAL TRIAL: NCT03046485
Title: A Randomized Controlled Trial to Assess if Attending an Interactive, Self-management Group, 'Living With Vision Loss', in Addition to Having Vision Rehabilitation in Our Clinic, Improves Patients' Quality of Life
Brief Title: Use of Self-management Group to Improve Quality of Life in Patients With Low Vision
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Mary Lou Jackson, principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-02-013; 07-02-013 (Other: Massachusetts Eye and Ear Center)
Record Dates: First submitted 2010-10-29; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; vision loss; self-management strategies; low-vision rehabilitation; IVI
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self management program (Experimental): Self management program 'Living with Vision Loss' 6 week course that met for 2 hours each week led by a trained leader.
  Interventions: Behavioral: Self management program 'Living with Vision Loss'
- Wait list control (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: Self management program 'Living with Vision Loss' — group met for 6 weeks, 2 hours per week, to discuss strategies for living with low vision
  Arms: Self management program

SUMMARY:
120 Patients with visual acuity <6/12 will be randomized to receive either usual care or participate in a 6-week, 2 hour 'Living with Vision Loss' program led by trained leaders. We hypothesize that a structured self-management low-vision rehabilitation program provides a greater improvement in participation in daily activities, and improves quality of life in vision-impaired people compared to the provision of the usual low vision rehabilitation services. We also plan to document barriers that prevent patients with low vision (visual acuity <6/12) from participating in self-management course.

ELIGIBILITY:
Inclusion Criteria:

* Clients who have attended the MEEI Vision Rehabilitation for the first time within 12 months
* Visual acuity of <6/12 in the better eye with habitual correction
* Age 55+ years
* Living independently (not in a nursing home)
* English speaking
* No cognitive impairment
* Adequate hearing to respond to normal conversation

Exclusion Criteria:

* vestibular disease

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Impact of Vision Impairment Questionnaire (IVI) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Jackson, MD, Principal Investigator — MEEI Vision REhabilitation Center Dir.
Locations (1):
- Vision Rehabilitation Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No